CLINICAL TRIAL: NCT04826497
Title: Effects of Nicorandil on Cardiac Sympathetic Nerve Activity and Distribution in Patients With Acute Myocardial Infarction Treated With Primary Percutaneous Coronary Intervention
Brief Title: Effect of Nicorandil on Cardiac Sympathetic Nerve for the Patients of Acute ST Segment Elevation Myocardial Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021KC20122
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Coronary Heart Disease
Keywords: nicorandil; primary percutaneous coronary intervention; acute ST segment elevation myocardial infarction; cardiac sympathetic nerve
MeSH Terms: conditions — Coronary Disease; ST Elevation Myocardial Infarction | interventions — Nicorandil; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicorandil (Experimental): Patients who received intracoronary and intravenous nicorandil before and after reperfusion with primary percutaneous coronary intervention
  Interventions: Drug: nicorandil
- Placebo （normal saline） (Placebo Comparator): Patients who received intracoronary and intravenous placebo before and after reperfusion with primary percutaneous coronary intervention
  Interventions: Drug: Placebo（normal saline）

INTERVENTIONS:
Drug: nicorandil — All patients received antiplatelet agents (aspirin, ticagrelor) and heparin.Diagnostic coronary angiography (CAG) was performed via the radial artery using the Seldinger method.The guidewire was passed into the culprit lesion.If the blood flow of culprit vessel reaches TIMI2-3 after balloon dilatation,6mg nicorandil was then administrated before stent implantation, A minimum 5-min interval occurred between the first and second doses of nicorandil to reduce adverse effects, subsequently , 6mg/h ivgtt. up to 48h after coronary intervention
  Other Names: Experiment Group
  Arms: Nicorandil
Drug: Placebo（normal saline） — All patients received antiplatelet agents (aspirin, ticagrelor) and heparin.Diagnostic coronary angiography (CAG) was performed via the radial artery using the Seldinger method.The guidewire was passed into the culprit lesion.If the blood flow of culprit vessel reaches TIMI2-3 after balloon dilatation,6mg placebo was then administrated before stent implantation, A minimum 5-min interval occurred between the first and second doses of placebo to reduce adverse effects, subsequently , 6mg/h ivgtt. up to 48h after coronary intervention
  Other Names: Control Group
  Arms: Placebo （normal saline）

SUMMARY:
The investigators evaluate the effects of intracoronary and intravenous administration of nicorandil on cardiac sympathetic nerve activity and distribution in patients with acute myocardial infarction undergoing primary percutaneous coronary intervention

DETAILED DESCRIPTION:
Reperfusion injury might occur in patients with acute ST segment elevation myocardial infarction undergoing the primary percutaneous coronary intervention(P-PCI),characterized by myocardial stunning, reperfusion-induced arrhythmia, microvascular dysfunction and injury of cardiac sympathetic nerve, etc.

Nicorandil is an antianginal agent with a dual mechanism of action: nitrate and K+ATP channel opener. The nitrate action causes vasodilation of systemic veins and epicardial coronary arteries, while the adenosine triphosphate (ATP)-sensitive potassium channel opener action causes vasodilation of peripheral and coronary resistance arterioles. Nicorandil not only decreases preload and afterload but also increases coronary blood flow.

The study will compare the effectiveness between nicorandil and placebo of preventing the reperfusion injury especially injury of cardiac sympathetic nerve in patients with acute ST segment elevation myocardial infarction undergoing the P-PCI.It is intended that before reperfusion injury ,nicorandil which was early used by intracoronary injection could prevent and release the microcirculatory spasm, release the coronary microvascular endothelial swelling,decrease embolism of atherosclerotic debris and thrombus formation,moreover,it could reduces the release of norepinephrine from sympathetic endings of the heart directly.So,it could decrease the phenomenon of no-reflow/slow reflow,reperfusion-induced arrhythmia and injury of cardiac sympathetic nerve.

ELIGIBILITY:
Inclusion Criteria:

1. acute ST-segment elevation myocardial infarction within 12 hours of symptom onset;
2. Age20-80,All genders
3. anterior myocardial infarction
4. The first myocardial infarction
5. The infarct-related artery(IRA) is totally occlusive
6. Blood pressure is higher than 90/60 millimeters of mercury（mmHg）
7. The time from myocardial infarction onset to reach the hospital is less than 12 hs

Exclusion Criteria:

1. kidney dysfunction (creatinine >2 mg/dl),
2. History of previous liver disease,
3. Cardiogenic shock,
4. History of myocardial infarction (MI)
5. History of coronary artery bypass grafting
6. History of allergic response to drugs
7. Severe hypovolemia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of the delayed heart/mediastinum count (H/M) ratio | 10 days after primary PCI
  The delayed heart/mediastinum count (H/M) ratio was determined from 123I-meta-iodobenzylguanidine (MIBG) images

SECONDARY OUTCOMES:
The total defect score (TDS) | 10 days after primary PCI
  The total defect score was determined from 123I-meta-iodobenzylguanidine (MIBG) images
Rate of slow re-flow/no-reflow phenomenon | 5 minutes after primary PCI
  TIMI myocardial perfusion grade (TMPG) of the final coronary flow in the culprit artery
Rate fo complete ST-segment resolution | 2 hours after primary PCI
  ST-segment resolution >50 percent in ECG
Rate of unplanned hospitalization for heart failure | 6 months after primary PCI
  Rate of unplanned hospitalization for heart failure
The washout rate (WR) | 10 days after primary PCI
  The washout rate (WR) were determined from 123I-meta-iodobenzylguanidine (MIBG) images
The total defect score (TDS) | 7 days after primary PCI
  The total defect score was determined from 99mTc-pyrophosphate scintigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Institute of Cardiovascular Disease Xuzhou Central Hospital, Study Director — Southeast University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Result] Piper HM, Meuter K, Schafer C. Cellular mechanisms of ischemia-reperfusion injury. Ann Thorac Surg. 2003 Feb;75(2):S644-8. doi: 10.1016/s0003-4975(02)04686-6. PMID 12607706
- [Result] Ji Z, Zhang R, Lu W, Ma G, Qu Y. The effect of nicorandil in patients with acute myocardial infarction undergoing percutaneous coronary intervention: a systematic review and meta-analysis. Ir J Med Sci. 2020 Feb;189(1):119-131. doi: 10.1007/s11845-019-02034-3. Epub 2019 May 30. PMID 31147987
- [Result] Xu L, Wang L, Li K, Zhang Z, Sun H, Yang X. Nicorandil prior to primary percutaneous coronary intervention improves clinical outcomes in patients with acute myocardial infarction: a meta-analysis of randomized controlled trials. Drug Des Devel Ther. 2019 Apr 29;13:1389-1400. doi: 10.2147/DDDT.S195918. eCollection 2019. PMID 31118574
- [Result] Fukui Y, Nozawa T, Ihori H, Sobajima M, Nakadate T, Matsuki A, Nonomura M, Fujii N, Inoue H, Kinugawa K. Nicorandil Attenuates Ischemia-Reperfusion Injury Via Inhibition of Norepinephrine Release From Cardiac Sympathetic Nerve Terminals. Int Heart J. 2017 Oct 21;58(5):787-793. doi: 10.1536/ihj.16-391. Epub 2017 Sep 30. PMID 28966311
- [Result] Kasama S, Toyama T, Kumakura H, Takayama Y, Ichikawa S, Suzuki T, Kurabayashi M. Effects of nicorandil on cardiac sympathetic nerve activity after reperfusion therapy in patients with first anterior acute myocardial infarction. Eur J Nucl Med Mol Imaging. 2005 Mar;32(3):322-8. doi: 10.1007/s00259-004-1672-0. Epub 2004 Oct 2. PMID 15791442
- [Result] Hicks KA, Mahaffey KW, Mehran R, Nissen SE, Wiviott SD, Dunn B, Solomon SD, Marler JR, Teerlink JR, Farb A, Morrow DA, Targum SL, Sila CA, Thanh Hai MT, Jaff MR, Joffe HV, Cutlip DE, Desai AS, Lewis EF, Gibson CM, Landray MJ, Lincoff AM, White CJ, Brooks SS, Rosenfield K, Domanski MJ, Lansky AJ, McMurray JJV, Tcheng JE, Steinhubl SR, Burton P, Mauri L, O'Connor CM, Pfeffer MA, Hung HMJ, Stockbridge NL, Chaitman BR, Temple RJ; Standardized Data Collection for Cardiovascular Trials Initiative (SCTI). 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials. J Am Coll Cardiol. 2018 Mar 6;71(9):1021-1034. doi: 10.1016/j.jacc.2017.12.048. PMID 29495982